CLINICAL TRIAL: NCT04486547
Title: Interviewing Adolescents With Type 1 Diabetes
Brief Title: Information Motivation Behavioral Skills Model's Effects on Adolescents With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elif Bakır (Other)
Responsible Party: Sponsor-Investigator, Elif Bakır, DR. Principal Investigator, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-059
Record Dates: First submitted 2020-07-08; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; adolescent; information motivation behavioral skills model,; nurse
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Follow up Posttest and HbA1c (No Intervention): 56.0% of the adolescents with type 1 diabetes were aged 12-14 years and 52.0% were male in the control group (n=25)
- Information Motivation Behavioral Skills Based Intervention (Experimental): 52.0% of the adolescents with type 1 diabetes were aged 15-18 years and 52.0% were female(n=25)
  Interventions: Behavioral: Information-Motivation-Behavioral Skills model-based intervention

INTERVENTIONS:
Behavioral: Information-Motivation-Behavioral Skills model-based intervention — Home visits were made to the study group and nursing interventions were administered in accordance with the components of the Information-Motivation-Behavioral Skills model
  Arms: Information Motivation Behavioral Skills Based Intervention

SUMMARY:
Aim: To evaluate the effects of information-motivation-behavioral skills model interventions given by nurses during home visits on the knowledge levels, personal and social motivation levels, behavioral skills, and HbA1C levels of adolescents with poor glycemic control.

Design: Randomized controlled study. Methods: 50 adolescents with type 1 diabetes were equally divided into study and control groups. Socio-Demographic Form, Diabetes Information Evaluation Form, The Child Attitude Toward Illness Scale, The Multidimensional Scale of Perceived Social Support, and Diabetes Management Self-Efficacy Scale were utilized in data collection. The scales were administered at the beginning of the study and six months later. HbA1c levels of adolescents were evaluated in the third and sixth months. Multiple home visits and phone calls were made to each participant in the intervention group. Interventions to improve the information-motivation-behavioral skills model-based knowledge, personal and social motivation, and behavioral skills were applied during the home visits.

DETAILED DESCRIPTION:
Aims The aim of the study was to evaluate the effects of IMB model interventions conducted by nurses during home visits on the knowledge levels, personal and social motivation levels, behavioral skills, and HbA1c levels of adolescents with T1DM. The study also aimed to test the following hypotheses: T1DM adolescents who experienced an IMB model-based intervention during a home visit will have more knowledge (H1) and more positive attitudes (H2) about their disease, higher levels of perceived social support (H3), higher levels of self-efficacy (H4), and lower levels of HbA1c (H5) than the control group Design A randomized controlled experimental study was conducted to test the hypotheses above and explore the aforementioned aim.

Sample/Participants The study was conducted with patients (n=50) of the Pediatric Endocrine Clinic of the Ankara Pediatric Hematology Oncology Training and Research Hospital between October 2018 and August 2019. The researchers evaluated the results of T1DM adolescents with HbA1c measurements at the clinic for 4 months and included those who met the inclusion criteria. The inclusion criteria were: (1) a T1DM diagnosis established at least six months ago, (2) an HbA1c level of >7.5, (3) not using insulin pumps, (4) the absence of any chronic disease other than diabetes, (5) attending follow-up visits at the clinic once every three months, and (6) living in Ankara. Adolescents were included in the study after an assessment of the HbA1c level. Adolescents who met the inclusion criteria were then grouped into study (n=25) and control (n=25) groups in order of arrival at the clinic, using stratified randomization by gender to ensure homogeneity.

The sample size was calculated based on the mean HbA1c level and standard deviations in the two groups in the power analysis made at the end of the research. An independent sample t-test was used to establish the 1.4-unit difference in mean HbA1c levels, and a power of 99.107% was achieved.

Data Collection The Sociodemographic Information Form prepared by the researcher consisted of six items regarding sociodemographic data and information on the participants.

Diabetes Information Evaluation Form (DIEF), Child Attitude toward Illness Scale (CATIS), Multidimensional Scale of Perceived Social Support (MSPSS), and Diabetes Management Self-Efficacy Scale (DMSES) were used to evaluate the components of the IMB model, and on the assessment of HbA1c.

The researcher attended a two-stage "Motivational Interviewing Techniques" course and received a certificate recognizing their ability to apply motivational interviewing techniques. The eligible participants and their parents were informed about the research, and written consent from the parents and written approvals from the adolescents were obtained.

Afterwards, home visits were made to the study group and nursing interventions were administered in accordance with the components of the IMB model. Information was provided in accordance with the adolescent's requirements, established from a pretest using the Diabetes Information Evaluation Form. For the personal motivation component, a list of obstacles and risky behaviors perceived by the patient in managing diabetes was created collaboratively. Patients were asked to think about the factors facilitating the emergence of such behaviors, as well as obstacles and negative perceptions, and potential solutions. Thereby, it aimed to raise the awareness of their risky behaviors. Furthermore, the patients were enabled to create positive values about themselves through the discovery of their strengths and weaknesses. As for social motivation, patients were supported in obtaining help from their loved ones when they felt unhappy. Cooperation with the diabetes team (physician, nurse, dietician) regarding appropriate topics was emphasized.

The skills of adolescents in activities such as blood glucose measurement, ketone measurement, insulin injection, record-keeping, administering additional insulin doses when required, creating a balanced food list, calculating the carbohydrate content of foods, and adjusting pre- and post-exercise insulin doses and meals were then evaluated. Feedback was provided enabling adolescents to correct their mistakes and improve self-efficacy.

During phone interviews, blood glucose results of the patient were determined first before the reasons were discussed. Taking into account the patient requirements, information was provided on insulin administration, nutrition, and exercise. The duration of the phone interviews varied from 2 to 15 minutes.

The control group adolescents received no intervention by the researcher throughout the study. For these participants, blood glucose measurement records were reviewed during their routine follow-ups at the hospital, their insulin doses were changed when necessary, and the daily intake of carbohydrates were adjusted after consultation with a dietician. The control group was informed that the scales would be re-administered six months later, and that they had to attend the hospital for HbA1c assessment at three and six months. After the posttest, incorrect answers by the control group were identified and information related to the question was provided.

Ethical Aspects of the Research Ethics committee approval was granted by the Health Sciences University Ankara Pediatric Hematology Oncology HARC Clinical Researches Ethics Committee on April 16, 2018 with case no: 2018-059.

Data Analysis Data were evaluated using IBM SPSS Statistics 23 software and a p value of <0.05 was considered statistically significant. The results of a Shapiro-Wilk test indicated a normal distribution of data, and so parametric tests were preferred in the study.

A dependent samples t-test was used to analyze the time-base differences of numerical variables at two different time points, while a repeated measures variance of analysis was used to examine the time-base differences at more than two different time points. The difference in the mean scale scores of the two groups were analyzed using an independent-samples t-test, while a Pearson's correlation analysis was used to examine the association between the scales. The power analysis of the research was carried out using NCSS PASS (Power Analysis and Sample Size) 11 software.

Validity and Reliability A Cronbach's alpha reliability analysis was performed to test the reliability of the scales

ELIGIBILITY:
Inclusion Criteria:

* 12-18 age An HbA1c level of ≥7.5

Exclusion Criteria:

* Diagnosed within the last 6 months An HbA1c level of ˂7.5 Using insulin pumps Having chronic diseases other than diabetes Living in another city Declining to participate

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline knowledge level of adolescents at 6 months | immediately before intervention and immediately after intervention
  Information evaluated by Diabetes Information Evaluation Form.The total information score was calculated over 20 points, with 1 point given for correct answers and 0 points to missing or wrong answers.
Change from baseline personal motivation level of adolescents at 6 months | immediately before intervention and immediately after intervention
  Personal motivation evaluated by Child Attitude toward Illness Scale. The nine items of the Child Attitude toward Ilness Scale are rated on a 5-point Likert-type scale.
Change from baseline behavioral skills level of adolescents at 6 months | immediately before intervention and immediately after intervention
  Diabetes Management Self-Efficacy Scale were used to evaluate Behavioral Skills. The instrument includes 26 items rated from 1 (strongly agree) to 5 (strongly disagree). A higher score indicates a lower level of self-efficacy.
Change from baseline HbA1c levels of adolescents at 6 months | immediately before intervention, at month 3 and immediately after intervention
  Before intervention, at month 3 and after intervention HbA1c levels of adolescents were evaluated for glycemic control
Change from baseline social motivation level of adolescents at 6 months | immediately before intervention and immediately after intervention
  Social motivation evaluated by Multidimensional Scale of Perceived Social Support. The Multidimensional Scale of Perceived Social Support consists of 12 items and it is rated on a 7-point Likert-type scale.

CONTACTS AND LOCATIONS:
Overall Officials: HİCRAN ÇAVUŞOĞLU, Study Chair — HACETTEPE UNIVESİTY NURSING FACULTY; EDA MENGEN, Study Chair — Ankara Pediatric Hematology Oncology Training and Research Hospital
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The results of the research will be published in the scientific journal and shared with other researchers